CLINICAL TRIAL: NCT00854984
Title: Pilot Study of a Practice Nurse Supported Psychological Self-help Intervention for Patients With Diabetes or Coronary Heart Disease and Co-morbid Depression
Brief Title: Pilot Study of a Self-help Intervention for Depression in Patients With a Chronic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: University of Stirling (Other); Robert Gordon University (Other); University of Glasgow (Other); Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Dr Margaret Maxwell, University of Stirling
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CZH/4/462; MREC: 08/H0405/39
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Depression; Diabetes Mellitus Type 2; Coronary Heart Disease
Keywords: Depression; diabetes; Coronary heart disease; CBT; Cognitive behavioural therapy
MeSH Terms: conditions — Depression; Diabetes Mellitus, Type 2; Coronary Disease; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-help CBT (Experimental): A nurse supported self-help CBT intervention in addition to usual care.
  Interventions: Behavioral: Living Life to the Full
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Living Life to the Full — A nurse-supported, self-help, cognitive behavioural therapy with web, video and booklet formats.
  Other Names: Five Areas
  Arms: Self-help CBT

SUMMARY:
A feasibility pilot trial of the self-help, "Cognitive behavioural therapy" based "Living Life to the Full" Materials for use by patients with diabetes type 2 and / or coronary heart disease.

DETAILED DESCRIPTION:
Depressed mood is common in patients with chronic disease and physical disability. It adversely affects quality of life, adherence to treatment and clinical outcome. Depression is expensive to the person, their family, employers and society. Recent developments in the UK General Practitioners' Contract mean that patients with two chronic diseases (Coronary Heart Disease- CHD and Diabetes - DM) are routinely screened for depression using a simple screening tool. We propose a study using an existing self help intervention in the specific context of patients with mild to moderately severe depression identified in this way.

This RCT is the second phase of a 2 phase mixed methods study examining the feasibility of a Full RCT. The first involved focus group with patients and health practitioners.

ELIGIBILITY:
Inclusion Criteria:

* Have had a diagnosis of diabetes mellitus type 2 and / or coronary heart disease.
* Be aged 35 or over.
* Be attending a participating primary care practice.
* Have a depression severity scale rating indicating moderate to moderately severe depression, such as:Prime-MD-PHQ9 of 10-21; HADS-D of 8-15;BDI-2 of 23-44

Exclusion Criteria:

* Unable to provide informed consent to participate
* Already receiving psychological treatment for their depression
* Have commenced treatment with an SSRI within the past 8 weeks
* Likely to have difficulty communicating by telephone
* Likely to have difficulty completing the forms and questionnaires
* Have a serious physical disorder
* Have a serious mental disorder
* Express significant suicidal thoughts (PHQ9 or BDI-2 question 9 scoring >1)
* Took part in an earlier related focus group

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-03-13 (Actual); Primary Completion 2009-09-30 (Actual); Study Completion 2009-09-30 (Actual)

PRIMARY OUTCOMES:
The obstacles to providing access and support to a generic online self help computerised cognitive behavioural therapy (CBT) programme for such patients. | 13 weeks

SECONDARY OUTCOMES:
The proportion of patients would prefer or require a non-computerised treatment alternative to treatment (i.e. a book or DVD based form of the treatment). | 13 weeks
The uptake, satisfaction with and completion of the self help programme when promoted and supported by practice nurses. | 13 weeks
A change in depression (BDI-2), anxiety , social function (WASAS), quality of life (Euroqol 5D) or illness perception (IPQ-R) from participation in a self help programme. | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Maxwell, PhD, Principal Investigator — University of Stirling
Locations (2):
- United Kingdom (2):
  - Faculty of Health and Social Care, Garthdee Campus, Robert Gordon University, Aberdeen
  - Community Health Sciences, GP Section, University of Edinburgh, Edinburgh